CLINICAL TRIAL: NCT01015924
Title: Intramedullary Nailing Compared With Plate Fixation of Displaced Mid-clavicular Fractures. A Prospective Randomized Controlled Trial
Brief Title: Plate Osteosynthesis Versus ESIN of Displaced Midclavicular Fractures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Hendrik Frolich Fuglesang, Assistant Prof. Stein Erik Utvåg, MD, PhD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rek 1.2009.1196
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Clavicle Fractures
Keywords: clavicle; TEN; Plate osteosynthesis; displaced; ESIN; displaced midshaft clavicular fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elastic Stable Intramedullary Nailing (Active Comparator): Operative intervention with closed or open reduction and intramedullary stabilization of midshaft clavicle fractures
  Interventions: Procedure: plate osteosynthesis; Procedure: ESIN
- Plate osteosynthesis (Active Comparator): Open reduction and plate fixation of midshaft clavicle fractures
  Interventions: Procedure: plate osteosynthesis; Procedure: ESIN

INTERVENTIONS:
Procedure: plate osteosynthesis — Patients are operated upon within 3 w of the fracture
  Other Names: The standard plate i a precontoured LCP clavicle plate by Synthes
Procedure: ESIN — Elastiv stable intramedullary nailing
  Other Names: TEN, synthes

SUMMARY:
The purpose of this study is to compare two widely used operative techniques on displaced midshaft clavicular fractures. The hypothesis is that there is no difference in functional outcome.

DETAILED DESCRIPTION:
Clavicular fracture is one of the most common fractures, accounting for about 4 % of all fractures. Midshaft fractures account for approximately 80%. Traditionally, midshaft fractures have been thought to have a good prognosis even when substantially displaced, and most have been treated nonoperatively with a sling or a figure of eight bandage. Early studies by Neer and Rowe in the 60´s demonstrated a very low non-union rate, with av prevalence of 4 in a series of 566 patients, and 3 nonunions in 2235 in another. On this basis, the general view has been that the vast majority of even severely displaced midshaft fractures healed uneventfully, with a very low nonunion rate and a good functional result. Operative results reported on the other hand bad results, especially concerning the risk of infection. Recent studies, however, conclude differently, and suggest the outcomes of displaced fractures might not be as favourable as once thought. Hill showed in a series of 52 completely displaced midclavicular fractures a nonunion rate of 15% (8 of 52 patients) and 31% (16 of 52) of patients were not satisfied with the end result. This correlated with a shortening of more than 2 cm. In a prospective study of 222 patients by Nowak, 42% (93 of 222) were found to have persisting symptoms after 6 months wheras 15% were found to have nonunion. These symptoms seem to persist even after 9 - 10 years reporting 29 % of 208 patients having pain during activity and 9% pain at rest. 46% did not consider themselves fully recovered.

Similar result were found in a systemic review of 2144 fractures. 15.1 % (24 of 159) of nonoperative treated dislocated fractures resulted in nonuion, whereas 2,2% (10 of 460) and 2% (5 of 152) nonunions were found in fractures treated operatively with either plate or intramedullary pins. On this basis, it is becoming more evident that conservative treatment gives much inferior results compared to earlier reported results.

The operative approach to midclavicular fractures have traditionally been plate osteosynthesis or intramedullary nailing. Poigenfürst in 1992 showed in a series of 122 patients a low nonunion rate and good functional results after plating. Likewise, intramedullary nailing has been described as an alternative technique with good results. Kettler demonstrated en a series of 87 patients a good functional results union in 97,7 % ( 85 of 87) and no infections. Similar results were fond by Rehm in 2004, with one nonunion of 136 fractures treated and a constant score one year after implant removal of 97.

Operative treatment of displaced midclavicular fracture thus shows reliable good results compared to earlier reported results. In 2007, the Canadian Orthopedic Trauma Society published a prospective randomised controlled trial of 132 patients, randomised to either conservative treatment with a sling, or plate fixation. The operative group showed clear superiority in Constant and DASH scores, reduction in risk of developing non-union, earlier return to work. With intramedullary nailing using ESIN technique, Smekal et al demonstrated superior results in the operative group in a prospective randomised controlled trial of 60 patients. 30 patients were opereated with elastic stable intramedullary nailing, and 30 patients were randomised to conservative treatment with a sling. The operative group had fewer complications, shorter time to union and a better functional outcome.

It seems from the above, that it is reasonable to offer operative treatment to active adults with displaced fractures of the middle third of the clavicle due to the risk of developing a symptomatic non- or malunion. Both plate fixation and intramedullary nailing of displaced fractures are described as safe methods of operative treatment. To our knowledge, there has never been conducted a prospective randomised controlled trial that compares different forms of the former mentioned operative alternatives.

On this basis, we plan to contuct a prospective randomised controlled trial comparing operative plate fixation and intramedullary nailing with TEN.

ELIGIBILITY:
Inclusion Criteria:

1. 16 - 60 years of age
2. Dislplaced midshaft clavicular fractures with no cortical bone contact or shortening over 15 mm
3. Tenting/compromised skin
4. Axial malalignment over 30 degrees

Exclusion Criteria:

1. More than 4 weeks old fracture
2. Ipsilateral damage that will influence the recovery and scoring systems, ie. Rotator cuff injury/fracture
3. Pathological fracture
4. Neurovascular injury
5. Open fracture
6. Noncompliance
7. Congenital anomaly or bone disease
8. Ongoing infectious process around the incision site for plate osteosynthesis

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2009-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Functional outcome using DASH score | quick dash w 1 thru 6. DASH at 6, 12, 26, 52

SECONDARY OUTCOMES:
At each control, complication such as infection, thoracic outlet syndrome is evaluated | continuously, as well as w 6, 12, 26, 52
Constant score | evaluated 6w, 12w, 26w 52 w
SF 36 | 26 w and 52 w

CONTACTS AND LOCATIONS:
Overall Officials: Stein Erik Utvag, MD PhD, Study Director — University of Oslo
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway